CLINICAL TRIAL: NCT00429247
Title: A Pilot Randomized Phase II Study of Adjuvant Administration of Trastuzumab (HERCEPTIN) Versus Observation After the Completion of Adjuvant Chemotherapy and Radiotherapy in Patients With Stage I-III Breast Cancer Who Have Detectable Disseminated and/or Circulating Tumor Cells (DTCs and/or CTCs) in the Bone Marrow or/and the Peripheral Blood Before or/and After the Completion of Adjuvant Treatment
Brief Title: Randomized Trial With Trastuzumab Versus Observation in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: V.Georgoulias, University Hospital of Crete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/01.60
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2008-01

CONDITIONS: Breast Cancer
Keywords: Occult tumor cells; Micrometastatic cells; Cytokeratin-19; Trastuzumab; Completion of Adjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Her
  Interventions: Drug: Trastuzumab
- 2 (No Intervention): Follow up

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab,first administration at the dose of 8mg/Kg IV, subsequent administrations at the dose of 6mg/Kg IV,every 3 weeks for 6 cycles
  Other Names: Herceptin
  Arms: 1

SUMMARY:
Epithelial tumor cells can be detected in the bone marrow and/or the peripheral blood [disseminated and circulating tumor cells, (DTCs) and (CTCs) respectively] of otherwise metastases-free patients with early breast cancer. Several studies have shown that the presence of these cells is an independent factor associated with an increased incidence of early disease relapse and disease-related death. In almost 50% of the patients, adjuvant chemotherapy cannot eliminate these occult tumor cells and this is also associated with a higher probability of early relapse and death. In 60-70% of the patients, DTCs and/or CTCs express the HER2/c-neu molecule and one or two administrations of their monoclonal antibody trastuzumab (HERCEPTIN) could eliminate these cells for a period ranging from 3-12 months.

DETAILED DESCRIPTION:
This pilot trial will compare the efficacy of the anti-HER2/erb-B2 monoclonal antibody trastuzumab (HERCEPTIN) given after the completion of the standard adjuvant chemotherapy and radiotherapy versus observation in patients with stage I-III operable breast cancer who have detectable cytokeratin-19 (CK-19) mRNA-positive tumor cells in the bone marrow or the peripheral blood before and/or after the adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Performance status (World Health Organization [WHO]) < 3
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function ( creatinine < 2 mg/dl)
* Adequate cardiac function (left ventricular ejection fraction [LVEF] > 50%).
* Informed consent
* Histologically or cytologically confirmed breast adenocarcinoma
* Prior surgical excision of the primary breast tumor
* Prior completion of standard adjuvant chemotherapy and/or radiotherapy
* Locally advanced disease after the completion of neo-adjuvant chemotherapy, surgical excision and radiotherapy provided that there was no evidence of local or metastatic disease
* Absence of any clinical or laboratory evidence of metastatic disease
* Detection of CTCs and/or DTCs (when it could be feasible) before the initiation and/or after the completion of adjuvant chemotherapy and/or radiotherapy
* Expression of HER2/c-neu on the primary tumor is not mandatory

Exclusion Criteria:

* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Other concurrent uncontrolled illness
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or nursing
* Positive pregnancy test
* History of allergic reaction attributed to trastuzumab (HERCEPTIN)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Compare the disease-free interval of patients with early-stage breast cancer | 3 years

SECONDARY OUTCOMES:
Elimination of CK-19 mRNA-positive CTCs. | Assessment of CK-19 mRNA CTCs every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (1):
- University Hospital of Crete, Heraklion, Crete, Greece